CLINICAL TRIAL: NCT03637829
Title: Effect of Mid-morning Snacks on Cognitive Performance, Satiety, Food Intake, and Glycemic Response in Normal Weight Adults
Brief Title: Effect of Morning Snack on Cognitive Performance in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Ryerson-REB-2017-339
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Nutrition; Cognitive Change; Food Intake Control; Satiety
Keywords: Healthy adults; Cognitive performance; Chocolate; Food intake; Glycemic response

STUDY DESIGN:
Intervention Model Description: A random and within subject, repeated measures experiment to study the effect of chocolate on cognitive performance, subjective appetite, food intake, and glycemic response in normal weight adults.
Who Masked: Participant, Investigator
Masking Description: treatments are in individual packages labelled "A", "B" and "C". Study participants and investigators are blinded to the composition of the test treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): 250 mL of water
  Interventions: Other: Control
- White Chocolate (Active Comparator): White chocolate (40 g)
  Interventions: Other: White chocolate
- Dark chocolate 1 (Experimental): Dark chocolate (40 g)
  Interventions: Other: Dark chocolate 1
- Dark chocolate 2 (Experimental): Dark chocolate (46 g) possibly containing caffeine and/or theobromine
  Interventions: Other: Dark chocolate 2

INTERVENTIONS:
Other: Control — Water
  Arms: Control
Other: White chocolate — Experimental snack treatment
  Arms: White Chocolate
Other: Dark chocolate 1 — Experimental snack treatment
  Arms: Dark chocolate 1
Other: Dark chocolate 2 — Experimental snack treatment
  Arms: Dark chocolate 2

SUMMARY:
To characterize the effects of three chocolate snacks on cognitive performance, subjective appetite, food intake control, and glycemic response in normal weight adults.

DETAILED DESCRIPTION:
On 4 separate mornings, 7 days apart, 12 hours after an overnight fast, and 3 hours after a standardized breakfast of a cereal bar, orange juice and fruit cup, participants will consume isocaloric snacks of white chocolate, 2 types of dark chocolate or control (water), followed by an ad libitum pizza lunch 90 minutes later. Upon arrival, at baseline (0 minutes), participants will be asked to complete the motivation-to-eat, global vigor and subjective emotion visual analogue scales (VAS), a battery of cognitive performance tasks and have blood samples taken, as reported and validated in our previous studies. Over the 90 minute testing period, blood samples will be taken,the VAS questions will be completed and cognitive tasks will be completed. Cognitive performance assessments will include learning and memory, spatial memory, attention and processing speed, and executive functions. VAS measuring physical comfort is completed pre- and post-meal. Ad libitum food intake from a test meal will be measured.

ELIGIBILITY:
Inclusion Criteria:

* be between 18 and 35 years of age
* be healthy and have a have body mass index (BMI) between 18.5 and 24.9
* not be taking any medications, not smoking, and
* not have allergies to chocolate, dairy or gluten
* be tested during the early follicular phase of their menstrual cycle for women

Exclusion Criteria:

* anyone with food sensitivities or allergies to chocolate, dairy or gluten,
* smokers
* diabetic or overweight/obese individuals.
* Restrained eating habits, defined as scoring greater than 11 points on the eating habits questionnaire

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Verbal declarative memory | At 15 minutes
  One of six word lists composed of 15 words will be audio presented and participants will be asked to write them down. The word list will be presented 3 times and the participant will immediately write down words after each time the word list is presented. This test will take 5 minutes
Change from baseline spatial memory | At Baseline, 15, 45, and 75 minutes
  Assessed using a spatial pattern recognition test on the Membrain Application. There will be a grid of 9 boxes with circles randomly located inside each box. Participants will be asked to remember where circles are located in each box. This test is done 6 times at each time-point, with each test having different random locations of circles. Each test will take 20 seconds.
Change in verbal declarative memory from the 15 minute time-point | At 45 and 75 minutes
  Participants will be asked to recall and write down all the words from the word list presented at the 15 minute time-point. This test will take 2 minutes.
Change from baseline executive function | At Baseline, 15, 45, and 75 minutes
  Will be assessed the Stroop task via the Membrain application. Participants will be presented with a list of words presented in colors that match the word (congruent, the word 'red' presented in red) or colors that do not match the word (incongruent, the word 'red' presented in blue). Participants will be asked to identify the color of the word, not the word itself. The task is scored for the number of correct and incorrect colors identified, as well as total time to completion. This test will be at each time-point and will take 1 minute to complete.
Change from baseline working memory and executive function | At Baseline, 15, 45, and 75 minutes
  A random 3 digit number will appear on the screen of the Membrain Application and the participant will have to continually subtract 3 from this number. At each time-point, participants will also complete the same test, except will subtract 7 continuously. This is a 2 minute test.
Change from baseline attention and reaction time | At Baseline, 15, 45, and 75 minutes
  Using the Membrain Application, Aa continuous string of single digit numbers appear on the screen, one at a time (each appearing for about one second). After seeing three consecutive ascending odd numbers, participants click the 'odd' button. When they see three consecutive, ascending even numbers, they click the 'even' button. When they see the number "1", they click the 'tertiary' button. This test is 5 minutes in length.

SECONDARY OUTCOMES:
Change from baseline subjective average emotions | At Baseline, 15, 30, 45, 60, 75 and 90 minutes
  Measured using 100 point visual analogue scales. Participants mark on this line to describe their feelings.
Change from baseline global vigor | At Baseline, 15, 30, 45, 60, 75 and 90 minutes
  Measured using 100 point visual analogue scales. Participants mark on this line to describe their feelings.
Change from baseline subjective average appetite | At Baseline, 15, 30, 45, 60, 75 and 90 minutes
  Measured using 100 point visual analogue scales. Participants mark on this line to describe their feelings.
Change from baseline blood glucose concentration | At Baseline, 15, 30, 45, 60, 75 and 90 minutes
  Blood glucose concentration (mmol/L) will be measured in whole blood using YSI 2300 STAT PLUS (YSI Incorporated, Yellow Springs, OH)
Food intake | At 90 minutes
  After other measures at the 90 minute time-point, participants will have lunch and food intake will be determined by weighing the meal before and after serving. The net weight of the test meal will be converted to kilocalories

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- School of Nutrition, Ryerson University, Toronto, Ontario, Canada